CLINICAL TRIAL: NCT06683079
Title: Comparison of the Effects of Hydroxyethyl Starch and Ringer's Lactate on Blood Loss and Coagulation After Colorectal Surgery.
Brief Title: Comparison Between Colloids and Crystalloids on Coagulation and Blood Loss
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Usama Mohammed Rabie, Assistant Lecturer, Assiut University
Other Study IDs: colloids versus crystalloids
Record Dates: First submitted 2021-07-25; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- colloid group: recieve colloids as a maintenance intraoperative fluid .
- crystalloid group: recieve crystalloids as a maintenance intraoperative fluid .

SUMMARY:
Infusion of intravenous fluids is mandatory especially in major and prolonged surgeries. However, there is no available optimum ideal type of fluid nor a fixed amount suitable for transfusion but it must be individualized for every patient to minimize the side effects of fluids.

Ringer's lactate as an example of crystalloids, causes a transient hypercoagulable state after its infusion, disappears in less than 6 hours of infusion and the coagulation profile returns to its state before Ringer's.

Voluven (Hydroxyehthyl starch 130/0.4) a colloid causes a hypocoagulable state after its infusion, and its effect is prolonged to more than 6 hours after infusion.

The effects of hydroxyethyl starch are not dose-dependent, but they can be remarkable even with mild to moderate amount of blood dilution applying nearly a restrictive fluid transfusion strategy and a goal-directed fluid therapy mode.

The amount of needed crystalloids is much more than that of colloids to maintain patients hemodynamically stable.

DETAILED DESCRIPTION:
When considering the optimum fluid of choice to achieve hemodynamic stability and the least morbidity, colloids have a theoritical and intuitive advantage. Being composed of molecules >35 kDa, colloids have traditionally been thought to have greater fluid efficacy (i.e. they remain in the intravascular space for longer ,thus contributing a greater effect on cardiac output) compared with crystalloids. These theoritical benefits of colloids led to their routine use in goal-directed therapy (GDT).

Studies in healthy volunteers have demonstrated that crystalloids tend to expand the intravascular volume by about 20% of the infused volume ;however when physiological endpoints have been used in clinical studies , the fluid efficacy of crystalloids increases up to 60%. This discrepancy may be explained by a number of factors, including the time taken for fluid to equilibrate throughout the extracellular fluid , the vaodilating effect of anethetic-indused hypotension on vascular capacitance, and the impairment of fluid elimination because of the surgical stress response.

While colloid has been the default fluid choice in most GDT studies to date, recent evidence from both the perioperative anesthestic setting and from intensive care have raised concerns that these agents may produce adverse effects on renal function and coagulation . recent studies have sought to compare the use of crystalloid solutions with colloids for GDT.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 to 75 years
* undergoing elective colorectal surgery

Exclusion Criteria:

* refusal by the patient
* patient with cardiac disease
* hepatic disease
* renal disease
* blood disease
* patient on regular anticoagulant drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient undergoing elective colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Prothrombin Time (PT) Measurement | Baseline just after induction, at end of infusion, and 6 hours post-operative.
  Measurement of Prothrombin Time to assess the effect of colloid and crystalloid administration on clotting time. Unit of Measure: seconds. Measurement Tool: laboratory tests were all supplied by technology of Marburg, Germany using Sysmex Cs 2100i, code (THL-02) with serial number 22880.
International Normalized Ratio (INR) | baseline just after induction, at end of infusion, 6 hours post-operative.
  Calculation of International Normalized Ratio to standardize clotting time measurements and evaluate the effect of fluid type on coagulation. Unit of Measure: ratio. Measurement Tool: laboratory tests were all supplied by technology of Marburg, Germany using Sysmex Cs 2100i, code (THL-02) with serial number 22880.
Activated Partial Thromboplastin Time (aPTT) | baseline just after induction, at end of infusion, 6 hours post-operative.
  Measurement of Activated Partial Thromboplastin Time to assess the intrinsic coagulation pathway after administration of colloid or crystalloid. Unit of Measure: seconds. Measurement Tool: laboratory tests were all supplied by technology of Marburg, Germany using Sysmex Cs 2100i, code (THL-02) with serial number 22880.
Factor V Levels | baseline just after induction, at end of infusion, 6 hours post-operative.
  Measurement of plasma levels of coagulation Factor V to evaluate changes in coagulation function following fluid administration. Unit of Measure: International Units per deciliter (IU/dL). Measurement Tool: laboratory tests were all supplied by technology of Marburg, Germany using Sysmex Cs 2100i, code (THL-02) with serial number 22880.
Factor VIII Levels | Baseline just after induction, at end of infusion, 6 hours post-operative.
  Plasma level measurement of coagulation Factor VIII to assess the impact of colloid and crystalloid on coagulation. Unit of Measure: International Units per deciliter (IU/dL). Measurement Tool: laboratory tests were all supplied by technology of Marburg, Germany using Sysmex Cs 2100i, code (THL-02) with serial number 22880.
Factor IX Levels | Baseline just after induction, at end of infusion, 6 hours post-operative.
  Measurement of coagulation Factor IX levels in plasma to assess any changes in the clotting profile after fluid administration. Unit of Measure: International Units per deciliter (IU/dL). Measurement Tool: laboratory tests were all supplied by technology of Marburg, Germany using Sysmex Cs 2100i, code (THL-02) with serial number 22880.
Blood Loss Volume | Total volume recorded at the end of the surgical procedure.
  Measurement of total blood loss volume to compare the effects of colloid and crystalloid solutions on hemostasis. Blood loss is calculated using the method outlined by Choi et al. (2010), which includes the volume in suction (minus irrigation fluid), visible blood on the surgical field, and blood absorbed in surgical pads. Surgical pads are estimated by inspection, with fully soaked pads counted as 150 mL and half-soaked pads as 100 mL. Unit of Measure: milliliters (mL).

SECONDARY OUTCOMES:
Blood transfusion requirements | Total units required recorded at the end of the surgical procedure.
  Assessment of the need for blood transfusions following administration of colloid or crystalloid solutions, to evaluate the effect of each solution on blood loss and hemostasis. Unit of Measure: number of transfusion units administered.

CONTACTS AND LOCATIONS:
Overall Officials: Kilany Ali Abdelsalam, Principal Investigator — Supervisor
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No